CLINICAL TRIAL: NCT02642744
Title: Improving Coordination and Transitions of Care for Stroke Patients With an Attending Nurse: a Comparative Effectiveness Single Center Study Comparing Models of Nursing Care
Brief Title: Improving Coordination and Transitions of Care in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823366
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Results first posted 2023-11-08 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Models, Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attending nurse model (Other): The attending nurse model of in-hospital care delivery aims to improve patient understanding, shared decision making, medication adherence, and reduce early readmissions after discharge to improve quality of life. On the inpatient stroke unit, the attending nurse will take ownership of essential aspects of an individual stroke patient's care, education, and transition out of the hospital. To further contribute to the patient's plan of care, the attending nurse will be present on daily teaching rounds.
  Interventions: Other: Nursing care model
- Conventional inpatient nursing care (No Intervention): Standard of care nursing care patients receive while inpatient

INTERVENTIONS:
Other: Nursing care model — Subjects will be randomized into either the attending nursing model of care vs the standard nursing model
  Arms: Attending nurse model

SUMMARY:
This study will examine if the attending nurse model will enhance critical patient-centered elements of care that will in turn improve patient education and shared decision-making, medication adherence, stroke-related health literacy, and reduce early readmissions to ultimately yield improved patient quality of life. Our primary objective is to determine whether the attending nurse model of care improves stroke patients' health at 7 days, 30 days, and 90 days after hospital discharge as assessed through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Admission to the Hospital of the University of Pennsylvania Vascular Neurology service
* Incident or recurrent:
* Ischemic stroke: focal neurological deficit of likely ischemic vascular origin
* Intracerebral hemorrhage: blood seen on initial head CT
* Transient Ischemic attack: focal neurological deficit of likely ischemic vascular origin that has clinically resolved

Exclusion Criteria:

* Pregnancy
* Comfort or hospice care
* Severe dementia prior to stroke
* Non-communicative and have no family/social support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-30 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Kasner, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attending Nurse Model | Conventional Inpatient Nursing Care
Started | 278 | 392
Completed | 129 | 169
Not Completed | 149 | 223

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attending Nurse Model | Conventional Inpatient Nursing Care | Total
Number analyzed (Participants) | 129 | 169 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (15) | 63 (16) | 63 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 78 | 132
  Male | 75 | 91 | 166
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 51 | 74 | 125
  White, Hispanic | 2 | 3 | 5
  African American, Non-Hispanic | 57 | 57 | 114
  Asian | 2 | 5 | 7
  Other | 16 | 23 | 39
  Missing | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 129 | 169 | 298

OUTCOME MEASURES:

1. Primary Outcome: Stroke Patient Education Retention Tool
Description: measures patient knowledge about stroke
Time Frame: 90 days
Population: These numbers reflect the number of participants that completed the measure
Measure: Count of Participants; unit: Participants
Arm/Group | Attending Nurse Model | Conventional Inpatient Nursing Care
Number analyzed (Participants) | 78 | 90
Participants
  Good | 49 | 52
  Bad | 29 | 38

2. Primary Outcome: Medication Compliance
Description: medication adherence measurement
Time Frame: 90 Days
Population: These numbers reflect the number of participants that completed the measure
Measure: Count of Participants; unit: Participants
Arm/Group | Attending Nurse Model | Conventional Inpatient Nursing Care
Number analyzed (Participants) | 82 | 94
Participants
  Adherent | 53 | 67
  Non-adherent | 29 | 27

ADVERSE EVENTS:
Time Frame: Up to 90 days after admission
Arm/Group | Attending Nurse Model | Conventional Inpatient Nursing Care
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/169
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/169
Other Adverse Events (participants affected / at risk) | 0/129 | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02642744/Prot_SAP_000.pdf